CLINICAL TRIAL: NCT03029988
Title: An Exploratory Evaluation of Technetium Tc 99m Tilmanocept by Intravenous (IV) Injection in Subjects With Liver Metastases From Colorectal Carcinoma Patients Using SPECT/CT Imaging Compared to Fluorodeoxyglucose (FDG) PET/CT Imaging.
Brief Title: An Evaluation of Tilmanocept by IV Injection Using SPECT/CT vs PET Imaging in Subjects With Liver Metastases.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of effect in Cohort 1
Sponsor: Navidea Biopharmaceuticals (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV3-25; 1R44CA162783-01 (NIH)
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Results first posted 2019-11-18 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Liver Metastases; Colorectal Carcinoma
Keywords: adenocarcinoma, Colorectal Carcinoma, liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Adenocarcinoma | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Intervention Model Description: Injection and imaging will begin with Cohort 1. Cohort 1 and Cohort 2 will receive tilmanocept intravenously.
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Subjects will receive 50 µg tilmanocept radiolabeled with 2.0 millicuries (mCi) Tc99m through a single IV injection.
  Interventions: Drug: Tilmanocept (Technetium Tc 99m tilmanocept Injection); Procedure: SPECT/CT Imaging
- Cohort 2 (Experimental): Subjects will receive 200 µg tilmanocept radiolabeled with 2.0 mCi Tc99m through a single IV injection.
  If it was determined that additional enrollment would not provide meaningful data, for example no metastatic liver lesions were visualized by Tc 99m tilmanocept for any of the subjects in the cohort, enrollment into Cohort 2 would begin and 3 subjects would be enrolled followed by a review of the imaging and safety data.
  Interventions: Drug: Tilmanocept (Technetium Tc 99m tilmanocept Injection); Procedure: SPECT/CT Imaging

INTERVENTIONS:
Drug: Tilmanocept (Technetium Tc 99m tilmanocept Injection) — Drug: Technetium Tc 99m tilmanocept
  Other Names: Lymphoseek
Procedure: SPECT/CT Imaging — 4-6 hours post-injection SPECT/CT will be obtained in the abdominal region.

SUMMARY:
Estimation of the concordance of Tc 99m localization in liver metastases from colorectal carcinoma using SPECT/CT imaging and abdominal FDG (PET)/CT imaging per subject.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-center, comparator study of IV injected Tc 99m Tilmanocept in the localization and detection of liver metastases in subjects with confirmed colorectal carcinoma (CRC). The study will be divided into two cohorts.

If it was determined that additional enrollment would not provide meaningful data, for example no metastatic liver lesions were visualized by Tc 99m tilmanocept for any of the subjects in the cohort, enrollment into Cohort 2 would begin and 3 subjects would be enrolled followed by a review of the imaging and safety data.

This study is designed to evaluate the safety and tolerability of Tc 99m tilmanocept administered intravenously. SPECT/CT imaging of the subject's abdominal cavity will be reviewed to establish concordance with FDG PET imaging.

ELIGIBILITY:
Inclusion Criteria:

* The subject has provided written informed consent with Health Information Portability and Accountability Act (HIPAA) authorization before the initiation of any study-related procedures.
* Subjects must be ≥18 years old;
* The subject must have a diagnosis of adenocarcinoma of the colon and/or rectum with FDG PET/CT confirmed metastases to the liver;
* The subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-3;
* The subject must be at least 4 weeks past any major intraabdominal surgery, including surgery to the liver;
* Subjects with prior malignancies other than colon and/or rectum cancer are allowed, provided they have been treated with curative intent, and have no evidence of recurrence of that malignancy;
* Each subject must have no more than 10 qualifying liver lesions that have been clinically confirmed metastatic adenocarcinoma of the colon by FDG PET/CT imaging.
* If of childbearing potential, the subject has a negative urine pregnancy test within 48 hours before administration of Tc 99m Tilmanocept, has been surgically sterilized, or has been postmenopausal for at least 1 year

Exclusion Criteria:

* The subject is pregnant or lactating.
* The subject has undergone any liver surgery, exclusive of a biopsy.
* The subject has known sensitivity to dextran.
* The subject has had preoperative chemotherapy, immunotherapy, or radiation therapy within the 10 days prior to Tc 99m Tilmanocept administration
* Before the administration of Tc 99m Tilmanocept, has received any radiopharmaceutical within 7 radioactive half-lives of that radiopharmaceutical
* Has received an investigational product within the 30 days prior to Tc 99m Tilmanocept administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick O Cope, PhD, Principal Investigator — Navidea Biopharmaceuticals
Locations (1):
- University of Alabama Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No subjects enrolled in Cohort 2
Groups:
- Cohort 1: Subjects will receive 50 µg tilmanocept radiolabeled with 2.0 mCi Tc99m through a single IV injection.
  Tilmanocept (Technetium Tc 99m tilmanocept Injection): Drug: Technetium Tc 99m tilmanocept
  SPECT/CT Imaging: 4-6 hours post-injection SPECT/CT will be obtained in the abdominal region.
Arm/Group | Cohort 1
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (16.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Visualization of Lesions by FDG PET/CT Imaging and by Tc 99m Tilmanocept SPECT/CT Imaging.
Description: The primary objectives of this study were to estimate the concordance of Tc 99m tilmanocept localization in liver metastases from colorectal carcinoma (CRC) using single photon emission computed tomography / computed tomography (SPECT/CT) imaging and abdominal fluorodeoxyglucose positron emission tomography-computed tomography (FDG PET/CT) imaging per subject and to evaluate the safety including monitoring the incidence of adverse events and changes over time in laboratory tests, vital signs, and physical examination findings.
Time Frame: Within 7 days after Tc 99m tilmanocept administration
Measure: Number; unit: Lesions
Groups:
- Cohort 1 - FDG PET CT: At screening, an FDG PET/CT scan was done in accordance with standard procedures
- Cohort 1 - Tilmanocept SPECT/CT: Subjects received 50 µg tilmanocept radiolabeled with 2.0 mCi Tc 99m through a single IV injection. SPECT/CT imaging of the abdominal region occurred 4-6 hours post-injection.
  Note: The liver lesion visualized by FDG PET/CT was excised prior to SPECT/CT imaging.
Arm/Group | Cohort 1 - FDG PET CT | Cohort 1 - Tilmanocept SPECT/CT
Number analyzed (Participants) | 3 | 3
Lesions
  Liver | 7 | 0
  Colon | 1 | 0

ADVERSE EVENTS:
Time Frame: 35 days
Arm/Group | Cohort 1
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) — Subject 25-01-005 experienced an adverse event (AE) of leukocytosis during their Follow-Up Visit laboratory evaluations
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) — Subject 25-01-002 reported an AE of hives after the Tc 99m tilmanocept administration (Visit 2, Day 1).

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and make modifications to the publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/88/NCT03029988/Prot_SAP_001.pdf